CLINICAL TRIAL: NCT00837187
Title: Bioavailability of Dexmedetomidine After Intranasal Administration in Healthy Subjects
Brief Title: Bioavailability of Dexmedetomidine After Intranasal Administration
Acronym: INDEX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Timo Iirola, Turku University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: INDEX
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Sedation
Keywords: dexmedetomidine; intranasal; pharmacokinetics; pharmacodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous dexmedetomidine (Active Comparator): Dexmedetomidine is administered intravenously
  Interventions: Drug: Intravenous dexmedetomidine
- Intranasal administration (Experimental): Dexmedetomidine is administered intranasally
  Interventions: Drug: Intranasal dexmedetomidine

INTERVENTIONS:
Drug: Intravenous dexmedetomidine — 100 ug
  Arms: Intravenous dexmedetomidine
Drug: Intranasal dexmedetomidine — 100 ug
  Arms: Intranasal administration

SUMMARY:
In a recent study by Yuen et al it was shown that preoperative intranasal administration of dexmedetomidine is a useful alternative for oral midazolam in children. However, there is no information on the pharmacokinetics of dexmedetomidine after intranasal administration.

The aim of this study is to investigate the comparative pharmacokinetics of intranasally and intravenously administered dexmedetomidine in healthy volunteers. The absolute bioavailability of intranasally administered dexmedetomidine will be calculated. In addition, we will report the effects of intranasally and intravenously administered dexmedetomidine on plasma catecholamine levels, systemic blood pressure, heart rate and sedation. We will also monitor the local and systemic safety and tolerability of intranasally administered dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* Fluent skills in the Finnish language in order to be able to give informed consent and communicate with the study personnel.
* Age ≥ 18 years.
* Male gender.
* Weight ≥ 60 kg.
* Written informed consent from the subject.

Exclusion Criteria:

* Previous history of intolerance to the study drug or related compounds and additives.
* Concomitant drug therapy of any kind except paracetamol in the 14 days prior to the study.
* Existing or recent significant disease.
* History of hematological, endocrine, metabolic or gastrointestinal disease.
* History of asthma or any kind of drug allergy.
* Previous or present alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements.
* Donation of blood within six weeks prior to and during the study.
* Special diet or lifestyle factors which would compromise the conditions of the study or the interpretation of the results.
* BMI > 30 kg / m2.
* Participation in any other clinical study involving investigational or marketed drug products concomitantly or within one month prior to the entry into this study.
* Smoking during one month before the start of the study or during the study period.
* Clinically significant abnormal findings in physical examination, ECG or laboratory screening [routine haematology (haemoglobin, haematocrit, red blood cell count, white blood cell count, platelets), renal function tests (creatinine, urea) and liver function tests (bilirubin)].

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The absolute bioavailability of intranasally administered dexmedetomidine | At baseline and 5, 10, 15, 20, 30, 45 min and 1, 1.5, 2, 3, 4, 5, 6, 8 and 10 h.

SECONDARY OUTCOMES:
The effects of intranasally and intravenously administered dexmedetomidine on plasma catecholamine levels, systemic blood pressure, heart rate and sedation, local and systemic safety and tolerability of intranasal dexmedetomidine. | At baseline and 5, 10, 15, 20, 30, 45 min and 1, 1.5, 2, 3, 5 and 10 h. Only local nasal tolerability is assessed at 5 and 10 h.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Iirola, MD, Principal Investigator — Turku University Hospital; Klaus T Olkkola, MD, PhD, Professor, Study Director — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Iirola T, Vilo S, Manner T, Aantaa R, Lahtinen M, Scheinin M, Olkkola KT. Bioavailability of dexmedetomidine after intranasal administration. Eur J Clin Pharmacol. 2011 Aug;67(8):825-31. doi: 10.1007/s00228-011-1002-y. Epub 2011 Feb 12. PMID 21318594